CLINICAL TRIAL: NCT00729079
Title: Virtual Translation of Diabetes Prevention to Primary Care: A Pilot Study
Brief Title: Diabetes Prevention Program Pilot Study
Acronym: DPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Geoffrey Williams, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24895
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Prevention
Keywords: Diabetes Prevention; Pre-Diabetes; Exercise; Fat Intake; Fasting blood sugar; tobacco cessation
MeSH Terms: conditions — Glucose Intolerance; Motor Activity; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subject will be randomly assigned to work with providers at Clinton Medical Associates
  Interventions: Behavioral: DPP
- 2 (Active Comparator): Subjects will be randomly assigned to work with providers at 1655 Elmwood AVe, Suite 125
  Interventions: Behavioral: DPP

INTERVENTIONS:
Behavioral: DPP — 1. The primary outcome measure is weight loss with a goal of 7% of initial weight.
  2. Secondary outcomes are adherence to behavior changes:
     1. Exercising a minimum of 150 minutes per week at a moderate level to maintain an energy expenditure of 700 kcals per week
     2. Fat intake less than 25% and saturated fat less than 10%
     3. Fiber intake of at least 25 grams per day
     4. Fasting blood sugar < 100 mg/dL
     5. Absence of tobacco use
  Arms: 1
Behavioral: DPP — 1. The primary outcome measure is weight loss with a goal of 7% of initial weight.
  2. Secondary outcomes are adherence to behavior changes:
     1. Exercising a minimum of 150 minutes per week at a moderate level to maintain an energy expenditure of 700 kcals per week
     2. Fat intake less than 25% and saturated fat less than 10%
     3. Fiber intake of at least 25 grams per day
     4. Fasting blood sugar < 100 mg/dL
     5. Absence of tobacco use
  Arms: 2

SUMMARY:
This pilot study is intended to demonstrate that we can actually deliver the Diabetes Prevention Program intervention well and to show that it is likely effective. We will use results from this pilot study to support our application to The National Institute of Health. NIH is asking for health care centers to show ways to provide this treatment at a reasonable cost. We propose to demonstrate successful and sustainable use DPP's lifestyle intervention in a primary care health care setting (University of Rochester Primary Care).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* BMI >24 kg/m2 (>22 kg/m2 among Asian Americans)
* IGT (2-h plasma glucose 140~199 mg/dl based on 75-g OGTT if available). The OGTT will not be required for inclusion, but the CMA practitioners may wish to recommend the OGTT for their patients.
* Elevated FPG (95~125 mg/dl*).
* HDL-triglyceride ration > 3.5.

Exclusion Criteria:

* Diabetes at baseline
* FPG >126 mg/dl*
* 2-h plasma glucose >200 mg/dl based on 75-g OGTT, if available. OGTT will not be required (see above note).
* Diabetes diagnosed by a physician and confirmed by other clinical data, other than during pregnancy.
* Ever used antidiabetic medication, other than during pregnancy
* Medical conditions likely to limit life span and/or increase risk of intervention
* Cardiovascular disease
* Hospitalization for treatment of heart disease in past 6 months New York Heart Association Functional Class> 2
* Left bundle branch block or third degree AV block Aortic stenosis
* Systolic blood pressure> 180 mmHg or diastolic blood pressure> 105 mmHg
* Cancer requiring treatment in the past 5 years, unless the prognosis is considered good
* Renal disease (creatinine GFR < or = 30 ml/hr or > 2.0 mg/dl if GFR not available).
* Anemia (hematocrit <36% in men or <33% in women)
* Hepatitis (based on history or serum transaminase elevation)
* Other gastrointestinal disease (pancreatitis, acute inflammatory bowel disease)
* Recent or significant abdominal surgery
* Pulmonary disease with dependence on oxygen or daily use of bronchodilators
* Chronic infection (e.g., HIV, active tuberculosis)
* Conditions or behaviors likely to affect conduct of the trial
* Unable to communicate with clinic staff (e.g., read and speak English).
* Unwilling to accept treatment assignment by randomization
* Participation in another intervention research project that might interfere with DPP
* Weight loss of > 10% in past 6 months for any reason except postpartum weight loss
* Unable to walk 0.25 miles in 10 min
* Currently pregnant or within 3 months postpartum
* Currently nursing or within 6 weeks of having completed nursing
* Pregnancy anticipated during the course of the trial
* Unwilling to undergo pregnancy testing or report possible pregnancy promptly
* Unwilling to take adequate contraceptive measures, if potentially fertile
* Major psychiatric disorder, including severe active major depression, severe anxiety, schizophrenia, manic depression, bi-polar disorder
* Excessive alcohol intake, either acute or chronic
* Medications and medical conditions likely to confound the assessment for diabetes including:

  * Niacin, in doses indicated for lowering serum triglycerides
  * Glucocorticoids, systemic
* Other prescription weight-loss medications
* Active Thyroid disease, suboptimally treated as indicated by abnormal serum thyroid-stimulating hormone
* Other endocrine disorders (e.g., Cushing's syndrome, acromegaly)
* Fasting plasma triglyceride >600 mg/dl, despite treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is weight loss with a goal of 7% of initial weight. | 6 months

SECONDARY OUTCOMES:
Exercising a minimum of 150 minutes per week at a moderate level to maintain an energy expenditure of 700 kcals per week | 6 months
;Fat intake less than 25% and saturated fat less than 10% Fiber intake of at least 25 grams per day;Fasting blood sugar < 100 mg/dL; Absence of tobacco use | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Williams, MD, PhD, Principal Investigator — University ofRochester; Heather Patrick, PhD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Clinton Medical Associated, Rochester, New York
  - Therapeutic Lifestyle Changes, Rochester, New York

REFERENCES:
- [Background] American Diabetes Association. Standards of medical care in diabetes--2008. Diabetes Care. 2008 Jan;31 Suppl 1:S12-54. doi: 10.2337/dc08-S012. No abstract available. PMID 18165335
- [Background] Benjamin SM, Valdez R, Geiss LS, Rolka DB, Narayan KM. Estimated number of adults with prediabetes in the US in 2000: opportunities for prevention. Diabetes Care. 2003 Mar;26(3):645-9. doi: 10.2337/diacare.26.3.645. PMID 12610015
- [Background] Goldstein MG, Whitlock EP, DePue J; Planning Committee of the Addressing Multiple Behavioral Risk Factors in Primary Care Project. Multiple behavioral risk factor interventions in primary care. Summary of research evidence. Am J Prev Med. 2004 Aug;27(2 Suppl):61-79. doi: 10.1016/j.amepre.2004.04.023. PMID 15275675
- [Background] Herman WH, Hoerger TJ, Brandle M, Hicks K, Sorensen S, Zhang P, Hamman RF, Ackermann RT, Engelgau MM, Ratner RE; Diabetes Prevention Program Research Group. The cost-effectiveness of lifestyle modification or metformin in preventing type 2 diabetes in adults with impaired glucose tolerance. Ann Intern Med. 2005 Mar 1;142(5):323-32. doi: 10.7326/0003-4819-142-5-200503010-00007. PMID 15738451
- [Background] Maciosek MV, Edwards NM, Coffield AB, Flottemesch TJ, Nelson WW, Goodman MJ, Solberg LI. Priorities among effective clinical preventive services: methods. Am J Prev Med. 2006 Jul;31(1):90-6. doi: 10.1016/j.amepre.2006.03.011. PMID 16777547
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Westfall JM, Mold J, Fagnan L. Practice-based research--"Blue Highways" on the NIH roadmap. JAMA. 2007 Jan 24;297(4):403-6. doi: 10.1001/jama.297.4.403. No abstract available. PMID 17244837
- [Background] Williams GC, Grow VM, Freedman ZR, Ryan RM, Deci EL. Motivational predictors of weight loss and weight-loss maintenance. J Pers Soc Psychol. 1996 Jan;70(1):115-26. doi: 10.1037//0022-3514.70.1.115. PMID 8558405
- See also: Diabetes Prevention Program — http://www.bsc.gwu.edu/dpp/manuals.htmlvdoc